CLINICAL TRIAL: NCT02454751
Title: The Use of Intranasal Fentanyl for the Treatment of Incident Dyspnea in Congestive Heart Failure: A Prospective Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Dr. Jana Pilkey, Physician, St. Boniface Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTA/2014/002
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Dyspnea; Congestive Heart Failure
MeSH Terms: conditions — Dyspnea; Heart Failure | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre-fentanyl dose/fentanyl dose (Experimental): Crossover: 6-six minute walk test, subjective rating of dyspnea, heart rate, respiratory rate, oxygen saturation and participants' general appearance measured before and after a dose of fentanyl.
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: fentanyl — One time dose of 50mcg of fentanyl administered intranasally
  Other Names: sublimaze

SUMMARY:
Study Objective The primary object of this study is to investigate the safety and effectiveness of fentanyl on the management of incident dyspnea.

Study Design The study design will be a cross over study with a minimum of a one hour wash out period.

DETAILED DESCRIPTION:
Clinical question and hypothesis In patients with congestive heart failure who experience episodic activity-induced dyspnea (incident dyspnea), will the administration of intranasal fentanyl pre-activity result in subjective improvement in dyspnea and objective improvement in functional capacity? Will there be side effects from this treatment?

We expect that pre-activity treatment with intranasal fentanyl will result in both subjective improvements in dyspnea ratings as well as an increased measurement of functional capacity. We also suspect that this treatment will not increase the patient's experienced side effects.

Study Objective The primary object of this study is to investigate the safety and effectiveness of fentanyl on the management of incident dyspnea.

Study Design The study design will be a cross over study with a minimum of a one hour wash out period.

Participation in this study will be for 2 hours over 1-2 days.

Primary Endpoints

• Walking distance from the 6MWT

Secondary Endpoints

* Subjective rating of dyspnea and side effects
* Heart rate, respiratory rate, oxygen saturation and participants' general appearance.

Sample Size We hope to study 20 patients. Given the paucity of data so far, it is not possible to statistically calculate the appropriate power for this study and 20 patients is an approximation based on clinical experience.

There is not enough data available currently for our statistician to find a power calculation that eliminates type 1 and 2 error. Based on anecdotal evidence and experience with this medication in the clinical setting, we have estimated that the number needed to determine a clinically relevant difference is likely around 20.

Patient Population We will study the application of fentanyl in patients ages 18 or older, of either gender, with either a diagnosis of NYHA Class 3 or 4 heart failure.

Inclusion Criteria

* Patients must be experiencing activity-induced incident dyspnea without reversible causes. They would have controlled background dyspnea without opioids.
* Patients must be physically able to safely ambulate in order to complete the 6MWT (may have mobility devices and may use supplement oxygen prescribed pre-study).

Exclusion Criteria

* Patients who are unable to perform the 6MWT for any reason or have contraindications to performing the 6MWT
* Patients that have anatomical pathologies that would make intranasal administration impossible
* Patients with known allergies/sensitivities to fentanyl/sufentanil

Withdrawal Criteria Participants may voluntarily withdraw from the study at any time they feel uncomfortable with the protocol. They will also be withdrawn if they experience chest pain, palpitations, syncope, presyncope, or worsening dyspnea. Objectively, they will be withdrawn if blood pressure drops below 90/50, heart rate drops below 60 or rises above 100, if oxygen saturation drops below 90%, or if respiratory rate drops below 8 or rises above 20. If any of: oxygen saturation, blood pressure, or respiratory rate drop below the cut off point and do not recover within 5 min of rest, the antidote, Naloxone will be administered with a subcutaneous injection. The trial may be stopped early if the treatment arm statistically demonstrates superiority or increased harm.

Treatment of Subjects All patients will do the walk test with and without and fentanyl. They will be instructed to continue any current medications that have been previously prescribed and to not make any changes to their medications. Should they be on any medications for dyspnea such as diuretics, bronchodilators, inhaled steroids, continuous oxygen, opioids etc., they are to be continued.

Before the first walk test, the patient will be asked to rate their baseline dyspnea, somnolence, anxiety, pain and nausea using the ESAS VAS scale. The research team will record baseline heart rate, respiratory rate, oxygen saturation and describe the patient's general appearance. The patient will complete the 6MWT under appropriate supervision from our research team.

The research team will re-measure the study patient's heart rate, respiratory rate, oxygen saturation and describe their general appearance for comparison to baseline. Any other adverse effects or symptoms will be recorded. These measures will be repeated at 10 minutes and 20 minutes post-6MWT to document any resolution of symptoms post activity. Following the 6MWT, treatment for dyspnea will be provided if required. The patient will also rerate their dyspnea, somnolence, anxiety, pain and nausea using the ESAS VAS scale for an objective measure.

After a minimum of 1 hour (wash out period), they will proceed to the second phase of the test.

For the second phase, the patient will once again be asked to rate their baseline dyspnea, somnolence, anxiety pain and nausea using the ESAS VAS scale. This is to ensure consistency among their baseline measures. The research team will record their objective measures as stated above. The patients will then be given the fentanyl treatment and the 6MWT will be repeated.

Patients would be administered a spray of 50mcg of fentanyl intranasally as suggested as the first titration step outlined in the Incident Pain and Dyspnea protocol, developed by the Winnipeg Regional Health Authority Palliative Care Program (http://palliative.info/IncidentPain.htm).

Following the 6MWT, the patient will again be asked to rate their baseline dyspnea, somnolence, anxiety and nausea using the ESAS VAS scale. The research team will complete and record objective measurements. As in phase 1 these measures will be repeated at 10 minutes and 20 minutes post-6MWT to document any resolution of symptoms post activity.

Assessment of Efficacy By collecting data at the time points described above, we will be able to compare the averaged baseline symptoms with exertion induced symptoms. Most importantly, the data will allow us to compare the difference in subjective symptoms between pre-exertional treatment with intranasal fentanyl with symptoms without pre-exertional treatment. Using the 6MWT, we would be able to objectively assess any change in the study patient's walking distance, which would represent a change in their functional capacity.

Assessment of Safety Patients will be monitored with a subjective symptom assessment scale (ESAS) and also with vital sign monitoring. If adverse events occur, the patients will be monitored by the research nurse with vitals signs taken every 5 minutes until the patient settles. If the patient does not settle within 5 minutes, as evidenced by an improvement in vital signs and/or subjective report, the research nurse will determine whether naloxone should be administered. If naloxone is not indicated, or the patient does not improve with the administration of naloxone, the research nurse will report the patient's condition to the patients primary nurse in charge of his/her care on the ward. The research nurse will further assist the primary nurse in providing standard medical care to the participant as necessary. If naloxone is administered, the research nurse will inform the primary ward nurse and will continue to monitor the patient with vital signs every 5 min for an hour. After an hour has elapsed, it is anticipated the study medication will have cleared from the participants body, and any unresolved adverse effects will be managed according to standard medical practice by the ward doctors and nurses. All adverse events will be documented. All serious adverse events (representing a significant health hazard to the participant) will be reviewed by the medical monitor and reported to the sponsor and the University of Manitoba Research Ethics Board and Health Canada accordingly.

Statistical Analysis Comparison of subjective rank data (non-parametric) between phase 1 and phase 2 will be analyzed using the Wilcoxin rank sum test. Comparison of objective numerical data (parametric) between phase 1 and 2 will be analyzed using paired t-tests. The 6MWT interpretation will include both absolute differences and percentage differences.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be experiencing activity-induced incident dyspnea without reversible causes. They would have controlled background dyspnea without opioids.
* Patients must be physically able to safely ambulate in order to complete the 6MWT (may have mobility devices and may use supplement oxygen prescribed pre-study).

Exclusion Criteria:

* Patients who are unable to perform the 6MWT for any reason or have contraindications to performing the 6MWT
* Patients that have anatomical pathologies that would make intranasal administration impossible
* Patients with known allergies/sensitivities to fentanyl/sufentanil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Walking distance from the 6MWT | 6 min
  meters walked

SECONDARY OUTCOMES:
Subjective rating of dyspnea and side effects (Edmonton Symptom Assessment Scale) | Day 1 - at time 0, 10 and 20 min Day 2 - at time 0, 10 and 20 min
  Edmonton Symptom Assessment Scale
respiratory rate | Day 1 - at time 0, 10 and 20 min Day 2 - at time 0, 10 and 20 min
  respirations in 1 minute
heart rate | Day 1 - at time 0, 10 and 20 min Day 2 - at time 0, 10 and 20 min
  heart beats in 1 minute
oxygen saturation | Day 1 - at time 0, 10 and 20 min Day 2 - at time 0, 10 and 20 min
  oxygen saturation as determined by oxygen saturation monitor
blood pressure | Day 1 - at time 0, 10 and 20 min Day 2 - at time 0, 10 and 20 min
  mmHg
general appearance (nurses subjective description) | Day 1 - at time 0, 10 and 20 min Day 2 - at time 0, 10 and 20 min
  nurses subjective description of patient dyspnea, color, sweating and voiced or unvoiced expressions of distress

CONTACTS AND LOCATIONS:
Overall Officials: Jana Pilkey, MD, Principal Investigator — St. Boniface Hosptial
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada